CLINICAL TRIAL: NCT04902677
Title: Relationship Between Parental Perception of Child's Weight and Feeding Practices in the Context of Childhood Obesity: The PERCEPS Study
Brief Title: Parental Perception of Child's Weight and Childhood Obesity
Acronym: PERCEPS
Status: Completed | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Sponsor
Other Study IDs: PERCEPS
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Childhood Obesity; Diet Habit
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- School
  Interventions: Other: Cross-sectional

INTERVENTIONS:
Other: Cross-sectional — No intervention

SUMMARY:
The increasing prevalence of metabolic diseases requires new strategies in the treatment and prevention of obesity. Children exposed to a poor diet and a sedentary lifestyle are especially vulnerable and may therefore be at risk of obesity at a very early stage in their lives. Recent studies have indicated a notable misperception of children's weight by parents. The main objective of this project is to study the association between parental perception of child's body weight and 1) feeding practices (permissive, restrictive or model); and 2) child's degree of overweight.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate

Exclusion Criteria:

-

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population consists in children from the 22 schools in the Sant Boi municipality (Barcleona, Spain). There are 5000 children of age beween 4-8 in these schools.
Sampling Method: Non-Probability Sample
Enrollment: 1898 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Infant feeding practices measured by the Child Feeding Practice questionnaire | Baseline
  We will assess three factors from the Child Feeding Practice (CFP) questionnaire measuring parental control practices and attitudes regarding child feeding: Restriction (8 items), Pressure to eat (4 items), and monitoring (3 items). Each item is scored from 1 to 5, and the mean value for each factor will be calculated.

SECONDARY OUTCOMES:
Participant BMI z-score | Baseline
  Weight and height of participants will be measured and combined to calculate the BMI z-score based on the WHO growth charts

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No